CLINICAL TRIAL: NCT06826248
Title: Clinical Efficacy of Darqeen Capsule for the Management of Hypothyroidism Associated with Female Reproductive Hormonal Imbalance
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Khadija Shaikh, M Phil Scholar, Hamdard University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-HLWP
Record Dates: First submitted 2025-02-01; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Female Infertility; Hormonal Imbalance; Qillat e Afraz e Darqiyya
MeSH Terms: conditions — Hypothyroidism; Infertility, Female

STUDY DESIGN:
Intervention Model Description: Single Blind, Single Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other)
  Interventions: Drug: Darqeen Capsule

INTERVENTIONS:
Drug: Darqeen Capsule — Effect of Darqeen capsule on Thyroid hormones

SUMMARY:
STUDY OBJECTIVES

1. To assess the safety of Darqeen capsule for the management of Hypothyroidism
2. Evaluate the efficacy of Darqeen capsule for the management of Hypothyroidism
3. To provide an alternative cost-effective treatment for the management of females suffering from hypothyroidism.

NULL HYPOTHESIS (HO) The Unani Medicine Darqeen capsule is not effective for the management of Hypothyroidism.

ALTERNATE HYPOTHESIS (H1) Unani medicine Darqeen capsule is effective for the management of Hypothyroidism.

DETAILED DESCRIPTION:
Hypothyroidism is a common endocrine disorder characterized by deficiency in the thyroid hormones, thyroxine (T4) and triiodothyronine (T3) which are crucial for regulating metabolism and maintaining overall bodily functions. There are several etiologies and manifestations of hypothyroidism. The most common clinical signs are weight gain, hair loss, sensitivity to cold, tiredness, constipation, dry skin, and voice changes.

The prevalence in Pakistan has been a growing concern, necessitating extensive research to address the underlying causes, risk factors, and optimal management strategies. It is estimated that hypothyroidism impacts approximately 5% of the population and 15% in females, with up to 5% possibly having undiagnosed thyroid failure. In Pakistan, the prevalence of hypothyroidism is reported to be 4.1%.

The description of Qillat-e-Ifraz-e-Darqiyya (hypothyroidism) in Unani system of medicine resembles the clinical manifestation associated with Su-e-Mizaj Barid Maddi (derangement in cold temperament).

The management of hypothyroidism involves thyroid hormone replacement therapy with levothyroxine, regular monitoring of hormone levels, and lifestyle modifications like a balanced diet, exercise, and stress management. Iodine supplementation is recommended in iodine-deficient regions, while underlying causes and pregnancy considerations should be managed. Educating patients about their condition and treatment plan is essential for active involvement in their health management.

Darqeen capsule is an Unani polyherbal formulation that primarily consists of natural ingredients, it is time tested pharmacopoeia formulation that is further modified by Hamdard Research Center. It is being used clinically for more than two years at Hamdard Matabs all around Pakistan and found effective for managing hypothyroidism and its associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with hypothyroidism
* Having raised TSH
* T3 & T4 hormones level below normal limits
* Females between the age group of 15-45 years

Exclusion Criteria:

* Subjects below the age group of 15 and above 45
* Suffering from chronic liver diseases and kidney failure, cancer or any other comorbid condition
* Currently taking any medication for Hypothyroidism or having history of adverse drug reaction
* Pregnant and lactating mothers.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Females
Enrollment: 50 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of TSH levels | 12 weeks
  Thyroid Stimulating Hormone-TSH level evaluated at baseline and compare with post treatment levels (after 12 weeks of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa Ul Mulk Memorial Hospital-Hamdard University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be share to ethical body